CLINICAL TRIAL: NCT04969562
Title: The Effect of Emotional Freedom Technique on Depressive Symptom, Anxiety and Psychological Distress of Individuals With New Diagnosis Multiple Sclerosis: A Randomized Controlled Study
Brief Title: The Effect of Emotional Freedom Technique on Depression, Anxiety and Distress of Individuals With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Neslihan Partlak Günüşen, Ass. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 6198-GOA
Record Dates: First submitted 2021-07-01; First posted 2021-07-20 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis; Anxiety; Depressive Symptoms; Psychiatric Nursing
Keywords: Multiple Sclerosis, anxiety, depression, pschological distress, emotional freedom technique
MeSH Terms: conditions — Multiple Sclerosis; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment (Experimental): Individuals with multiple sclerosis in the experimental group will be included in six sessions of EFT at seven-day intervals, in which one session lasts 30-45 minutes. SUDS will be applied before and after each EFT session. At the same time, resting heart rate and blood pressure will be measured in the EFT group before and after each session.
  Interventions: Behavioral: Emotional Freedom Technique
- control (No Intervention): They will continue their routine treatment.

INTERVENTIONS:
Behavioral: Emotional Freedom Technique — Emotional Freedom Technique (EFT, Emotional Freedom Technique) is a psychophysiological interpretation that combines elements of cognitive behavioral therapy (CBT), exposure therapy, and somatic stimulation using acupuncture points.
  Arms: experiment

SUMMARY:
Volunteers over the age of 18 who applied to the Neurology Outpatient Clinic of Dokuz Eylül University Hospital, who were diagnosed with multiple sclerosis in the last three months, one month after the initiation of treatment and accepted the study, will be included in the study after their eligibility to the sampling criteria is evaluated. EDSS will be applied to the individuals by the specialist physician and they will be directed to the MS daycare unit. Since it is a randomized controlled experimental study, the sampling and follow-up measurements will be carried out by a psychologist in the unit where the study is applied, who does not carry out EFT. Scales will be applied in the daily unit and will be randomly divided into two groups at the beginning of the study. The psychologist who chooses the sampling will not know which group the participants will fall into, and the EFT practitioner will not know the anxiety, depression and psychological distress levels of the individuals participating in the study. EFT will be applied to one of the groups, and the other group will continue their routine treatment. Individuals with multiple sclerosis in the experimental group seven days at intervals, six sessions in which one session lasts 30-45 minutes will be included in the EFT application. SUDS will be applied before and after each EFT session. At the same time, resting heart rate and blood pressure will be measured in the EFT group before and after each session. Depression, anxiety and psychological distress levels of individuals with MS will be evaluated with HAD and SUDS at the beginning of the study, at the end of six sessions and in the first month.

DETAILED DESCRIPTION:
Multiple sclerosis (MS); It is an autoimmune central nervous system (CNS) disease characterized by inflammation, demyelination and axon damage, progressing with attacks and remissions. It ranks first among the diseases that cause neurological disability in adults, regardless of trauma. Being diagnosed with MS usually creates a state of shock in patients and it takes time to get used to the disease. Individuals with MS have to struggle daily with various physical, cognitive and psychological symptoms such as walking and movement limitations, pain, fatigue, depression, memory and concentration difficulties. This type of chronic disease, which occurs in adulthood (between the ages of 20-40), increases the size of the problems because it is seen in a period when life is most active and functional, and family, social and professional goals and activities are at the highest level. Individuals with MS may be prone to depression and anxiety due to various psychosocial risk factors such as inadequate coping or inadequate social support, as well as biological processes associated with MS (such as changes in brain structure or immunological and inflammatory pathways). Psychiatric symptoms may occur before the diagnosis, when the first neurological symptoms appear, or after diagnosis as indicated in retrospective studies.

Because depression and anxiety can worsen over time in individuals with MS, it is important to improve early recognition and management of these symptoms. Individuals with MS experience intense anxiety and stress in the process from the first symptoms to the diagnosis process. Depression affects 15 to 47% of individuals with MS, and this rate is much higher than other chronic neurological diseases and is three times higher than in the general population. Anxiety disorders are present in 36-54% of the MS population, and approximately 30% of individuals with MS have symptoms consistent with generalized anxiety disorder. It is important to create short and cost-effective interventions to reduce depressive symptoms, psychological distress, and improve the quality of life of individuals with MS. Emotional Freedom Technique (EFT) is a psychophysiological intervention that combines elements of cognitive behavioral therapy (CBT), exposure therapy, and somatic stimulation using acupuncture points. EFT is an intervention in which one's physical or psychological awareness focuses on a specific issue and simultaneously stimulates selected acupuncture points along the body meridians, especially on the head and upper body, by touching them with the fingertips. Since it is a simple applicable, evidence-based self-help technique like EFT, it is a suitable first-line option for treating psychiatric symptoms. As a safe and reliable self-help method, EFT is highly effective in reducing symptoms of depression in a wide range of settings and demographic groups and shows clinical benefit as a low-cost drug-free treatment. It is also suggested that EFT improves symptoms occurring in more than one physiological system simultaneously.

Determining and intervening the depression or anxiety levels of individuals with MS is especially important in the treatment of newly diagnosed individuals. For these symptoms, EFT is a short, easy, reliable, cost-effective and self-administered method, while being a self-administered method allows the individual to manage the disease. The aim of this study is to examine the effect of EFT on depressive symptoms, anxiety, psychological distress levels, SDMT scores, resting heart rate and blood pressure in individuals with newly diagnosed multiple sclerosis.

The study will consist of volunteers over the age of 18 who have been diagnosed with multiple sclerosis in the last three months, one month has passed since the treatment was started, followed in the Neurology Outpatient Clinic of Dokuz Eylul University Medical Faculty Hospital or treated in the MS Day Treatment Unit. 50 participants, including 2 groups (with EFT and no EFT), will be included in the study. EDSS will be applied to individuals by a specialist physician. They will be referred to the MS day treatment unit. Since it is a randomized controlled experimental study, the sample and follow-up measurements will be carried out by a psychologist in the unit where the research is conducted, who does not carry out the EFT application. Scales will be applied in the daily unit. The study will be randomized and divided into two groups at the beginning. The psychologist who made the sampling selection will not know which group the participants will belong to, and the EFT practitioner will not know the anxiety, depression and psychological distress levels of the individuals participating in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Being over 18 years old
2. Being cooperative and oriented enough to follow the given instructions
3. Having been diagnosed with MS in the last three months
4. Having been on MS treatment for at least a month
5. Getting a score of 3 and above on the SUDS scale

Exclusion Criteria:

1. Being in the flare of psychiatric illness
2. Using psychiatric medication for less than three months
3. Having an MS attack

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline anxiety levels at 6 weeks assessed by anxiety subscale of Hospital Anxiety Depression Scale (HADS) | Change from Baseline Anxiety at 6 weeks
  In this study, Hospital Anxiety Depression Scale is used to determine the anxiety levels of individuals with MS. Consisting of 14 questions in total, the seven items measure the anxiety. The cut-off point is 10 for the anxiety.The minimum score that can be obtained from the anxiety sub-dimension of the scale is 0 and the maximum score is 21.
  The higher the score, the higher the anxiety level. Higher score mean a worse outcome.
Change from baseline depressive symptoms levels at 6 weeks assessed by depressive symptoms subscale of Hospital Anxiety Depression Scale (HADS) | Change from Baseline depressive symptoms at 6 weeks
  In this study, Hospital Anxiety Depression Scale is used to measure depressive symptoms of individuals with MS. Consisting of 14 questions in total, the seven measure the depressive symptoms. For subscale, 0-7 points were predicted to be the normal range, 8-10 points were predicted to be considered, and 11 points were predicted to be over-estimated mood.The minimum score that can be obtained from the depression sub-dimension of the scale is 0 and the maximum score is 21.
  The higher the score, the higher the depressive symptoms level.Higher score mean a worse outcome.
Change from baseline psychological distress symptoms levels at 6 weeks assessed by Subjective Units of Distress Scale (SUDS). | Change from Baseline distress at 6 weeks
  In this study, the Subjective Units of Distress Scale (SUDS) is used to assess the level of psychological distress. SUDS scores provide concrete and basic data about the individual's condition at the beginning and at the end of therapy, thus reflecting changes that may occur in the process. SUDS is frequently used by studies in the literature for the evaluation of EFT results. Participants typically identify a concern or problem they want to address and rate their level of distress on a Likert-type scale out of 10 (10 is the maximum amount of distress and 0 represents the minimum or neutral situation). By means of this scoring, the severity of the discomfort felt by the individual at that moment is determined. This figure serves as a concrete and basic starting point regarding the state of the individual at the time of implementation. Thus, at the end of the application, it gives the opportunity to obtain an indicator reflecting the change provided by the application.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No